CLINICAL TRIAL: NCT05292261
Title: Effects of a Short- and Long-term Team Handball-based Exercise Programme on Physical Fitness and Health Status of Inactive Postmenopausal Women
Brief Title: Effects of a Recreational Team Handball-based Programme on Health and Physical Fitness of Postmenopausal Women
Acronym: H4HW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Institute of Maia (Other)
Collaborators: Research Center in Sports Sciences, Health Sciences and Human Development (Other); Universidade do Porto (Other); Laboratory of Metabolism and Exercise (LaMetEx), CIAFEL, Faculty of Sport, University of Porto (Unknown); Centre of Research, Education, Innovation and Intervention in Sport, University of Porto (Unknown); University of Southern Denmark (Other); Porto Sports Medicine Center (IPDJ, IP) (Unknown); Gaia City Hall (Unknown); Portuguese Handball Federation (Unknown); European Handball Federation (Unknown); São João University Hospital Centre (Unknown); EPIUnit, Public Health Institute, University of Porto (Unknown)
Responsible Party: Principal Investigator, Susana Cristina Araújo Póvoas, Associate Professor, University Institute of Maia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CEFADE202019
Record Dates: First submitted 2022-03-14; First posted 2022-03-23 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Menopause

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Team handball group (Experimental): The team handball group participants were encouraged to performed at least two out of three weekly supervised team handball training sessions of 60 min each, for 36 weeks.
  Interventions: Other: Recreational team handball
- Control group (No Intervention): The control group participants were instructed to keep their regular daily physical activity for 36 weeks.

INTERVENTIONS:
Other: Recreational team handball — Two to three weekly sessions of recreational team handball training for 36 weeks. Each 60-min session started with a standardised warm-up (including running, coordination, strength, flexibility, and balance exercises) followed by three 15-min periods of recreational team handball matches, interspersed by 2-min breaks, played as small-sided games (4v4, 5v5 or 6v6). The training sessions were performed on an indoor team handball court (40x20 m) adjusted to result in 34-36 m2 per player. During the matches, the participants rotated positions every 3 min in a random order, including the goalkeeper and no exclusions or substitutions were applied.
  Arms: Team handball group

SUMMARY:
This study aimed at determining the short- (16 weeks) and long-term (36 weeks) health and physical fitness effects and adherence of recreational team handball training for postmenopausal women without previous experience with the sport.

The investigators hypothesized that short-term recreational team handball training would result in positive health and physical fitness adaptations and that the health and physical fitness improvements achieved after the first 16 weeks would be maintained or further improved at the long-term. Moreover, the investigators also hypothesized that the adherence to this exercise mode would be maintained throughout the 36 weeks (long-term) compared to the first 16 weeks (short-term).

ELIGIBILITY:
Inclusion Criteria:

* Inactive postmenopausal women aged +55 years or younger if with menopause for at least 3 years

Exclusion Criteria:

* Any medical contraindications to perform moderate-to-vigorous physical activity

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Postmenopausal women
Enrollment: 80 (Actual)
Dates: Start 2016-01-02 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Between group differences in peak oxygen uptake at week 16 | Week 16
  Determined by pulmonary gas exchange measurements, during an incremental treadmill test until voluntary exhaustion.
Between group differences in peak oxygen uptake at week 36 | Week 36
  Determined by pulmonary gas exchange measurements, during an incremental treadmill test until voluntary exhaustion.
Changes from baseline in peak oxygen uptake at week 16 | Baseline and week 16
  Determined by pulmonary gas exchange measurements, during an incremental treadmill test until voluntary exhaustion.
Changes from baseline in peak oxygen uptake at week 36 | Baseline and week 36
  Determined by pulmonary gas exchange measurements, during an incremental treadmill test until voluntary exhaustion.
Changes from week 16 in peak oxygen uptake at week 36 | Week 16 and week 36
  Determined by pulmonary gas exchange measurements, during an incremental treadmill test until voluntary exhaustion.

SECONDARY OUTCOMES:
Between group differences in resting heart rate at week 16 | Week 16
  Determined by an automatic upper arm blood pressure monitor according to standardized procedures.
Between group differences in resting heart rate at week 36 | Week 36
  Determined by an automatic upper arm blood pressure monitor according to standardized procedures.
Changes from baseline in resting heart rate at week 16 | Baseline and week 16
  Determined by an automatic upper arm blood pressure monitor according to standardized procedures.
Changes from baseline in resting heart rate at week 36 | Baseline and week 36
  Determined by an automatic upper arm blood pressure monitor according to standardized procedures.
Changes from week 16 in resting heart rate at week 36 | Week 16 and week 36
  Determined by an automatic upper arm blood pressure monitor according to standardized procedures.
Between group differences in body mass at week 16 | Week 16
  Determined by whole-body dual- energy X-ray absorptiometry following standard procedures.
Between group differences in body mass at week 36 | Week 36
  Determined by whole-body dual- energy X-ray absorptiometry following standard procedures.
Changes from baseline in body mass at week 16 | Baseline and week 16
  Determined by whole-body dual- energy X-ray absorptiometry following standard procedures.
Changes from baseline in body mass at week 36 | Baseline and week 36
  Determined by whole-body dual- energy X-ray absorptiometry following standard procedures.
Changes from week 16 in body mass at week 36 | Week 16 and week 36
  Determined by whole-body dual- energy X-ray absorptiometry following standard procedures.
Between group differences in fat mass at week 16 | Week 16
  Determined by whole-body dual- energy X-ray absorptiometry following standard procedures.
Between group differences in fat mass at week 36 | Week 36
  Determined by whole-body dual- energy X-ray absorptiometry following standard procedures.
Changes from baseline in fat mass at week 16 | Baseline and week 16
  Determined by whole-body dual- energy X-ray absorptiometry following standard procedures.
Changes from baseline in fat mass at week 36 | Baseline and week 36
  Determined by whole-body dual- energy X-ray absorptiometry following standard procedures.
Changes from week 16 in fat mass at week 36 | Week 16 and week 36
  Determined by whole-body dual- energy X-ray absorptiometry following standard procedures.
Between group differences in lean mass at week 16 | Week 16
  Determined by whole-body dual- energy X-ray absorptiometry following standard procedures.
Between group differences in lean mass at week 36 | Week 36
  Determined by whole-body dual- energy X-ray absorptiometry following standard procedures.
Changes from baseline in lean mass at week 16 | Baseline and week 16
  Determined by whole-body dual- energy X-ray absorptiometry following standard procedures.
Changes from baseline in lean mass at week 36 | Baseline and week 36
  Determined by whole-body dual- energy X-ray absorptiometry following standard procedures.
Changes from week 16 in lean mass at week 36 | Week 16 and week 36
  Determined by whole-body dual- energy X-ray absorptiometry following standard procedures.
Between group differences in lumbar spine bone mineral density at week 16 | Week 16
  Determined by dual- energy X-ray absorptiometry regional scans following standard procedures.
Between group differences in lumbar spine bone mineral density at week 36 | Week 36
  Determined by dual- energy X-ray absorptiometry regional scans following standard procedures.
Changes from baseline in lumbar spine bone mineral density at week 16 | Baseline and week 16
  Determined by dual- energy X-ray absorptiometry regional scans following standard procedures.
Changes from baseline in lumbar spine bone mineral density at week 36 | Baseline and week 36
  Determined by dual- energy X-ray absorptiometry regional scans following standard procedures.
Changes from week 16 in lumbar spine bone mineral density at week 36 | Week 16 and week 36
  Determined by dual- energy X-ray absorptiometry regional scans following standard procedures.
Between group differences in dominant femur bone mineral density at week 16 | Week 16
  Determined by dual- energy X-ray absorptiometry regional scans following standard procedures.
Between group differences in dominant femur bone mineral density at week 36 | Week 36
  Determined by dual- energy X-ray absorptiometry regional scans following standard procedures.
Changes from baseline in dominant femur bone mineral density at week 16 | Baseline and week 16
  Determined by dual- energy X-ray absorptiometry regional scans following standard procedures.
Changes from baseline in dominant femur bone mineral density at week 36 | Baseline and week 36
  Determined by dual- energy X-ray absorptiometry regional scans following standard procedures.
Changes from week 16 in dominant femur bone mineral density at week 36 | Week 16 and week 36
  Determined by dual- energy X-ray absorptiometry regional scans following standard procedures.
Between group differences in dominant femoral neck bone mineral density at week 16 | Week 16
  Determined by dual- energy X-ray absorptiometry regional scans following standard procedures.
Between group differences in dominant femoral neck bone mineral density at week 36 | Week 36
  Determined by dual- energy X-ray absorptiometry regional scans following standard procedures.
Changes from baseline in dominant femoral neck bone mineral density at week 16 | Baseline and week 16
  Determined by dual- energy X-ray absorptiometry regional scans following standard procedures.
Changes from baseline in dominant femoral neck bone mineral density at week 36 | Baseline and week 36
  Determined by dual- energy X-ray absorptiometry regional scans following standard procedures.
Changes from week 16 in dominant femoral neck bone mineral density at week 36 | Week 16 and week 36
  Determined by dual- energy X-ray absorptiometry regional scans following standard procedures.
Between group differences in lumbar spine bone mineral content at week 16 | Week 16
  Determined by dual- energy X-ray absorptiometry regional scans following standard procedures.
Between group differences in lumbar spine bone mineral content at week 36 | Week 36
  Determined by dual- energy X-ray absorptiometry regional scans following standard procedures.
Changes from baseline in lumbar spine bone mineral content at week 16 | Baseline and week 16
  Determined by dual- energy X-ray absorptiometry regional scans following standard procedures.
Changes from baseline in lumbar spine bone mineral content at week 36 | Baseline and week 36
  Determined by dual- energy X-ray absorptiometry regional scans following standard procedures.
Changes from week 16 in lumbar spine bone mineral content at week 36 | Week 16 and week 36
  Determined by dual- energy X-ray absorptiometry regional scans following standard procedures.
Between group differences in dominant femur bone mineral content at week 16 | Week 16
  Determined by dual- energy X-ray absorptiometry regional scans following standard procedures.
Between group differences in dominant femur bone mineral content at week 36 | Week 36
  Determined by dual- energy X-ray absorptiometry regional scans following standard procedures.
Changes from baseline in dominant femur bone mineral content at week 16 | Baseline and week 16
  Determined by dual- energy X-ray absorptiometry regional scans following standard procedures.
Changes from baseline in dominant femur bone mineral content at week 36 | Baseline and week 36
  Determined by dual- energy X-ray absorptiometry regional scans following standard procedures.
Changes from week 16 in dominant femur bone mineral content at week 36 | Week 16 and week 36
  Determined by dual- energy X-ray absorptiometry regional scans following standard procedures.
Between group differences in dominant femoral neck bone mineral content at week 16 | Week 16
  Determined by dual- energy X-ray absorptiometry regional scans following standard procedures.
Between group differences in dominant femoral neck bone mineral content at week 36 | Week 36
  Determined by dual- energy X-ray absorptiometry regional scans following standard procedures.
Changes from baseline in dominant femoral neck bone mineral content at week 16 | Baseline and week 16
  Determined by dual- energy X-ray absorptiometry regional scans following standard procedures.
Changes from baseline in dominant femoral neck bone mineral content at week 36 | Baseline and week 36
  Determined by dual- energy X-ray absorptiometry regional scans following standard procedures.
Changes from week 16 in dominant femoral neck bone mineral content at week 36 | Week 16 and week 36
  Determined by dual- energy X-ray absorptiometry regional scans following standard procedures.
Between group differences in osteocalcin at week 16 | Week 16
  Determined by chemiluminescence method using a fully automated immunoassay system.
Between group differences in osteocalcin at week 36 | Week 36
  Determined by chemiluminescence method using a fully automated immunoassay system.
Changes from baseline in osteocalcin at week 16 | Baseline and week 16
  Determined by chemiluminescence method using a fully automated immunoassay system.
Changes from baseline in osteocalcin at week 36 | Baseline and week 36
  Determined by chemiluminescence method using a fully automated immunoassay system.
Changes from week 16 in osteocalcin at week 36 | Week 16 and week 36
  Determined by chemiluminescence method using a fully automated immunoassay system.
Between group differences in procollagen type-1 amino-terminal propeptide at week 16 | Week 16
  Determined by chemiluminescence method using a fully automated immunoassay system.
Between group differences in procollagen type-1 amino-terminal propeptide at week 36 | Week 36
  Determined by chemiluminescence method using a fully automated immunoassay system.
Changes from baseline in procollagen type-1 amino-terminal propeptide at week 16 | Baseline and week 16
  Determined by chemiluminescence method using a fully automated immunoassay system.
Changes from baseline in procollagen type-1 amino-terminal propeptide at week 36 | Baseline and week 36
  Determined by chemiluminescence method using a fully automated immunoassay system.
Changes from week 16 in procollagen type-1 amino-terminal propeptide at week 36 | Week 16 and week 36
  Determined by chemiluminescence method using a fully automated immunoassay system.
Between group differences in carboxy-terminal type-1 collagen crosslinks at week 16 | Week 16
  Determined by chemiluminescence method using a fully automated immunoassay system.
Between group differences in carboxy-terminal type-1 collagen crosslinks at week 36 | Week 36
  Determined by chemiluminescence method using a fully automated immunoassay system.
Changes from baseline in carboxy-terminal type-1 collagen crosslinks at week 16 | Baseline and week 16
  Determined by chemiluminescence method using a fully automated immunoassay system.
Changes from baseline in carboxy-terminal type-1 collagen crosslinks at week 36 | Baseline and week 36
  Determined by chemiluminescence method using a fully automated immunoassay system.
Changes from week 16 in carboxy-terminal type-1 collagen crosslinks at week 36 | Week 16 and week 36
  Determined by chemiluminescence method using a fully automated immunoassay system.
Between group differences in sclerostin at week 16 | Week 16
  Determined by chemiluminescence method using a fully automated immunoassay system.
Between group differences in sclerostin at week 36 | Week 36
  Determined by chemiluminescence method using a fully automated immunoassay system.
Changes from baseline in sclerostin at week 16 | Baseline and week 16
  Determined by chemiluminescence method using a fully automated immunoassay system.
Changes from baseline in sclerostin at week 36 | Baseline and week 36
  Determined by chemiluminescence method using a fully automated immunoassay system.
Changes from week 16 in sclerostin at week 36 | Week 16 and week 36
  Determined by chemiluminescence method using a fully automated immunoassay system.
Between group differences in isometric knee extension peak torque at week 16 | Week 16
  Determined by a Biodex isokinetic dynamometer, during a isometric knee extension contraction
Between group differences in isometric knee extension peak torque at week 36 | Week 36
  Determined by a Biodex isokinetic dynamometer, during a isometric knee extension contraction
Changes from baseline in isometric knee extension peak torque at week 16 | Baseline and week 16
  Determined by a Biodex isokinetic dynamometer, during a isometric knee extension contraction
Changes from baseline in isometric knee extension peak torque at week 36 | Baseline and week 36
  Determined by a Biodex isokinetic dynamometer, during a isometric knee extension contraction
Changes from week 16 in isometric knee extension peak torque at week 36 | Week 16 and week 36
  Determined by a Biodex isokinetic dynamometer, during a isometric knee extension contraction
Between group differences in isometric knee extension rate of force development at week 16 | Week 16
  Determined by a Biodex isokinetic dynamometer, during a isometric knee extension contraction
Between group differences in isometric knee extension rate of force development at week 36 | Week 36
  Determined by a Biodex isokinetic dynamometer, during a isometric knee extension contraction
Changes from baseline in isometric knee extension rate of force development at week 16 | Baseline and week 16
  Determined by a Biodex isokinetic dynamometer, during a isometric knee extension contraction
Changes from baseline in isometric knee extension rate of force development at week 36 | Baseline and week 36
  Determined by a Biodex isokinetic dynamometer, during a isometric knee extension contraction
Changes from week 16 in isometric knee extension rate of force development at week 36 | Week 16 and week 36
  Determined by a Biodex isokinetic dynamometer, during a isometric knee extension contraction
Between group differences in upper body strength at week 16 | Week 16
  Determined by a handgrip dynamometer.
Between group differences in upper body strength at week 36 | Week 36
  Determined by a handgrip dynamometer.
Changes from baseline in upper body strength at week 16 | Baseline and week 16
  Determined by a handgrip dynamometer.
Changes from baseline in upper body strength at week 36 | Baseline and week 36
  Determined by a handgrip dynamometer.
Changes from week 16 in upper body strength at week 36 | Week 16 and week 36
  Determined by a handgrip dynamometer.
Between group differences in postural balance at week 16 | Week 16
  Determined by the number of falls in a single-legged flamingo balance test.
Between group differences in postural balance at week 36 | Week 36
  Determined by the number of falls in a single-legged flamingo balance test.
Changes from baseline in postural balance at week 16 | Baseline and week 16
  Determined by the number of falls in a single-legged flamingo balance test.
Changes from baseline in postural balance at week 36 | Baseline and week 36
  Determined by the number of falls in a single-legged flamingo balance test.
Changes from week 16 in postural balance at week 36 | Week 16 and week 36
  Determined by the number of falls in a single-legged flamingo balance test.
Between group differences in aerobic performance at week 16 | Week 16
  Determined by meters covered in the Yo-Yo intermittent endurance level 1 test.
Between group differences in aerobic performance at week 36 | Week 36
  Determined by meters covered in the Yo-Yo intermittent endurance level 1 test.
Changes from baseline in aerobic performance at week 16 | Baseline and week 16
  Determined by meters covered in the Yo-Yo intermittent endurance level 1 test.
Changes from baseline in aerobic performance at week 36 | Baseline and week 36
  Determined by meters covered in the Yo-Yo intermittent endurance level 1 test.
Changes from week 16 in aerobic performance at week 36 | Week 16 and week 36
  Determined by meters covered in the Yo-Yo intermittent endurance level 1 test.
Between group differences in total cholesterol at week 16 | Week 16
  Determined by an automated analyser.
Between group differences in total cholesterol at week 36 | Week 36
  Determined by an automated analyser.
Changes from baseline in total cholesterol at week 16 | Baseline and week 16
  Determined by an automated analyser.
Changes from baseline in total cholesterol at week 36 | Baseline and week 36
  Determined by an automated analyser.
Changes from week 16 in total cholesterol at week 36 | Week 16 and week 36
  Determined by an automated analyser.
Between group differences in high-density lipoprotein cholesterol at week 16 | Week 16
  Determined by an automated analyser.
Between group differences in high-density lipoprotein cholesterol at week 36 | Week 36
  Determined by an automated analyser.
Changes from baseline in high-density lipoprotein cholesterol at week 16 | Baseline and week 16
  Determined by an automated analyser.
Changes from baseline in high-density lipoprotein cholesterol at week 36 | Baseline and week 36
  Determined by an automated analyser.
Changes from week 16 in high-density lipoprotein cholesterol at week 36 | Week 16 and week 36
  Determined by an automated analyser.
Between group differences in low-density lipoprotein cholesterol at week 16 | Week 16
  Determined by an automated analyser.
Between group differences in low-density lipoprotein cholesterol at week 36 | Week 36
  Determined by an automated analyser.
Changes from baseline in low-density lipoprotein cholesterol at week 16 | Baseline and week 16
  Determined by an automated analyser.
Changes from baseline in low-density lipoprotein cholesterol at week 36 | Baseline and week 36
  Determined by an automated analyser.
Changes from week 16 in low-density lipoprotein cholesterol at week 36 | Week 16 and week 36
  Determined by an automated analyser.
Between group differences in triglycerides at week 16 | Week 16
  Determined by an automated analyser.
Between group differences in triglycerides at week 36 | Week 36
  Determined by an automated analyser.
Changes from baseline in triglycerides at week 16 | Baseline and week 16
  Determined by an automated analyser.
Changes from baseline in triglycerides at week 36 | Baseline and week 36
  Determined by an automated analyser.
Changes from week 16 in triglycerides at week 36 | Week 16 and week 36
  Determined by an automated analyser.
Between group differences in fasting glucose at week 16 | Week 16
  Determined by an automated analyser.
Between group differences in fasting glucose at week 36 | Week 36
  Determined by an automated analyser.
Changes from baseline in fasting glucose at week 16 | Baseline and week 16
  Determined by an automated analyser.
Changes from baseline in fasting glucose at week 36 | Baseline and week 36
  Determined by an automated analyser.
Changes from week 16 in fasting glucose at week 36 | Week 16 and week 36
  Determined by an automated analyser.
Between group differences in fasting insulin at week 16 | Week 16
  Determined by an automated analyser.
Between group differences in fasting insulin at week 36 | Week 36
  Determined by an automated analyser.
Change from baseline in fasting insulin at week 16 | Baseline and week 16
  Determined by an automated analyser.
Change from baseline in fasting insulin at week 36 | Baseline and week 36
  Determined by an automated analyser.
Change from week 16 in fasting insulin at week 36 | Week 16 and week 36
  Determined by an automated analyser.
Between group differences in glucose tolerance at week 16 | Week 16
  Determined by an oral glucose tolerance teste, analysed by an automated analyser.
Between group differences in glucose tolerance at week 36 | Week 36
  Determined by an oral glucose tolerance teste, analysed by an automated analyser.
Changes from baseline in glucose tolerance at week 16 | Baseline and week 16
  Determined by an oral glucose tolerance teste, analysed by an automated analyser.
Changes from baseline in glucose tolerance at week 36 | Baseline and week 36
  Determined by an oral glucose tolerance teste, analysed by an automated analyser.
Changes from week 16 in glucose tolerance at week 36 | Week 16 and week 36
  Determined by an oral glucose tolerance teste, analysed by an automated analyser.

CONTACTS AND LOCATIONS:
Overall Officials: Susana Póvoas, Principal Investigator — University of Maia
Locations (1):
- University of Maia, Maia, Porto District, Portugal